CLINICAL TRIAL: NCT04440033
Title: Factors Associated with Falling in Parkinson's Disease: a Multidisciplinary Prospective Study
Brief Title: Factors Associated with Falling in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: BC-07392
Record Dates: First submitted 2020-06-03; First posted 2020-06-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Accidental Falls; Risk factor; Gait; Speech; Audiology
MeSH Terms: conditions — Parkinson Disease; Speech

STUDY DESIGN:
Intervention Model Description: Case-control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parkinson's Disease group (Experimental): Patients with stage 3 idiopathic Parkinson's Disease
  Interventions: Other: Baseline assessment of demographic, anthropometric and clinical characteristics; Other: Locomotor assessments; Other: Speech assessments; Other: Audiology assessments
- Healthy control group (Active Comparator): Age and sex-matched healthy adults
  Interventions: Other: Baseline assessment of demographic, anthropometric and clinical characteristics; Other: Locomotor assessments; Other: Speech assessments; Other: Audiology assessments

INTERVENTIONS:
Other: Baseline assessment of demographic, anthropometric and clinical characteristics — * Age
  * Sex
  * Height
  * Body weight
  * Handedness
  * Medication use
  * Blood pressure
  * Global cognition (Montreal Cognitive Assessment)
  * Fear of falling (Shortened Iconographical Falls Efficacy Scale)
  * History of falls (number of falls in the past month)
  * Time since diagnosis and symptom onset
  * Disease severity (UPDRS part III, Hoehn and Yahr)
  * Non-motor symptoms (UPDRS part I)
  * Motor symptoms (UPDRS part III)
  * Motor complications (UPDRS part IV)
  * Disease-dominant side (UPDRS part III)
  * Freezing of gait (New Freezing of Gait Questionnaire)
  Arms: Parkinson's Disease group
Other: Baseline assessment of demographic, anthropometric and clinical characteristics — * Age
  * Sex
  * Height
  * Body weight
  * Handedness
  * Medication use
  * Blood pressure
  * Global cognition (Montreal Cognitive Assessment)
  * Fear of falling (Shortened Iconographical Falls Efficacy Scale)
  * History of falls (number of falls in the past month)
  Arms: Healthy control group
Other: Locomotor assessments — First, 9 anthropometric measurements will be taken, 39 reflective markers will be placed, and a 6-min practice walking session will be conducted to familiarize participants with self-paced treadmill walking (SPTW). Thereafter, participants will partake in 7 experimental conditions in a (semi-)randomized order:
  * 3 min standing
  * 3 min standing while answering semi-standardized questions
  * 3 min SPTW
  * 3 min SPTW while answering semi-standardized questions (SPTW-Q)
  * 3 min SPTW while verbally describing a VR environment (SPTW-VR1)
  * 6 min SPTW in a VR environment containing freezing of gait provoking elements (SPTW-VR2)
Other: Speech assessments — * Acoustic analysis (including voice reports and formant analysis), video recording and motor speech profile (including analysis of diadochokinesis, voice, standard syllabic rate, intonation and second formant (F2)).
  * Spontaneous speech production will be assessed by answering semi-standardized questions based on the Aachen Aphasia Test and by describing a VR environment projected on a 180-degree cylindrical screen
  * The Speech Handicap Index (a 15-item self-reported questionnaire)
Other: Audiology assessments — * Otoscopy
  * Tympanometry
  * Pure tone audiometry
  * Otoacoustic emissions
  * Video Head Impuls Test
  * Cervical Vestibular Evoked Myogenic Potentials
  * Ocular Vestibular Evoked Myogenic Potentials
  * Oculomotor function testing
  * Positional testing
  * Static visual acuity test
  * Dynamic visual acuity test
  * Dizziness Handicap Inventory (a 25-item self-assessment inventory)

SUMMARY:
The objective of this study will be to identify multidisciplinary fall risk factors in persons with stage 3 idiopathic Parkinson's Disease compared to age and sex-matched healthy adults. Both the relative contribution of each independent factor, as well as the interaction between these factors, will be examined. The study will include multidisciplinary assessments, including locomotor, speech, auditory, vestibular and opthalmologic assessments.

ELIGIBILITY:
Parkinson's Disease group

Inclusion criteria:

* Persons with idiopathic PD diagnosed by a medical doctor according to the United Kingdom PD Brain Bank Criteria
* Aged between 18 and 75 years-old
* Stage 3 on the Hoehn and Yahr scale in the on-medication state
* On a stable dose of PD medication (at least one week)
* Able to stand and walk on a treadmill without support for at least 3 minutes
* Able to give consent

Exclusion criteria:

* Atypical parkinsonism
* Unpredictable symptom fluctuations
* Previous surgical management of PD (i.e., deep brain stimulation surgery; pallidotomy)
* Duodopa pump therapy
* Dementia (Montreal Cognitive Assessment (MoCA) < 21)[1]
* Symptomatic orthostatic hypotension (e.g. frequent syncope episodes)
* Concurrent neurological disorders (e.g. stroke)
* Comorbidities that affect gait or balance (e.g. peripheral neuropathy)
* Acute illness
* Epilepsy or history of seizures
* Depression (MDS-UPDRS item 1.3 ≥ 2)
* Body weight over 120 kilograms
* Pregnancy
* Participation in other ongoing experimental trials

Healthy control group

Inclusion criteria:

* Age and sex-matched healthy adults

Exclusion criteria:

* Symptomatic orthostatic hypotension (e.g. frequent syncope episodes)
* Body weight over 120 kilograms
* Pregnancy
* Participation in other ongoing experimental trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Fall events | baseline to 6 months after baseline
  Number of accidental falls documented using a daily fall diary with monthly telephone follow-ups.

SECONDARY OUTCOMES:
Walking speed | baseline during 3 min self-paced treadmill walking; baseline during 3 min self-paced treadmill walking while answering semi-standardized questions; baseline during 3 min self-paced treadmill walking while describing a virtual environment
  Walking speed (meters/second) measured using the Gait Real-time Interactive Lab (GRAIL) system (Motekforce Link, The Netherlands).
Walking cadence | baseline during 3 min self-paced treadmill walking; baseline during 3 min self-paced treadmill walking while answering semi-standardized questions; baseline during 3 min self-paced treadmill walking while describing a virtual environment
  Walking cadence (steps/minute) measured using the Gait Real-time Interactive Lab (GRAIL) system (Motekforce Link, The Netherlands).
Step length | baseline during 3 min self-paced treadmill walking; baseline during 3 min self-paced treadmill walking while answering semi-standardized questions; baseline during 3 min self-paced treadmill walking while describing a virtual environment
  Step length (meters) measured using the Gait Real-time Interactive Lab (GRAIL) system (Motekforce Link, The Netherlands).
Hip, knee and ankle joint angle during walking | baseline during 3 min self-paced treadmill walking; baseline during 3 min self-paced treadmill walking while answering semi-standardized questions; baseline during 3 min self-paced treadmill walking while describing a virtual environment
  Hip, knee and ankle joint angle during walking (°) measured using the Gait Real-time Interactive Lab (GRAIL) system (Motekforce Link, The Netherlands).
Hip, knee and ankle joint moment during walking | baseline during 3 min self-paced treadmill walking; baseline during 3 min self-paced treadmill walking while answering semi-standardized questions; baseline during 3 min self-paced treadmill walking while describing a virtual environment
  Hip, knee and ankle joint moment during walking (Nm/kg) measured using the Gait Real-time Interactive Lab (GRAIL) system (Motekforce Link, The Netherlands).
Hip, knee and ankle joint power during walking | baseline during 3 min self-paced treadmill walking; baseline during 3 min self-paced treadmill walking while answering semi-standardized questions; baseline during 3 min self-paced treadmill walking while describing a virtual environment
  Hip, knee and ankle joint moment during power (W/kg) measured using the Gait Real-time Interactive Lab (GRAIL) system (Motekforce Link, The Netherlands).
Freezing of gait | baseline during 6 min self-paced treadmill walking in a virtual environment
  Number of freezing of gait events measured using the Gait Real-time Interactive Lab (GRAIL) system (Motekforce Link, The Netherlands).
Spontaneous speech production | baseline; baseline during 3 min self-paced treadmill walking; baseline during 3 min self-paced treadmill walking while answering semi-standardized questions; baseline during 3 min self-paced treadmill walking while describing a virtual environment
  Audio recordings analyzed using PRAAT software to assess spontaneous speech production
Spontaneous speech production | baseline; baseline during 3 min self-paced treadmill walking; baseline during 3 min self-paced treadmill walking while answering semi-standardized questions; baseline during 3 min self-paced treadmill walking while describing a virtual environment
  Audio recordings analyzed using Motor Speech Profile software to assess spontaneous speech production
Speech Handicap Index | baseline
  A 15-item self-reported questionnaire based on the Parole Handicap Index to evaluate the physical, functional and psychosocial impact of dysarthria (0-60). Higher scores indicate a higher level of speech-related problems.
Otoscopy | baseline
  A otoscopic test to examine the external auditory canal and the tympanic membrane
Tympanometry | baseline
  An auditory test to assess the middle-ear function
Pure tone audiometry | baseline
  An auditory test to assess hearing threshold levels
Otoacoustic Emissions Test | baseline
  An auditory test to measure cochlear outer hair cell function
Video Head Impuls Test | baseline
  A vestibular function test to objectify high frequency function of the horizontal and vertical semicircular canals
Cervical Vestibular Evoked Myogenic Potential Testing | baseline
  A vestibular function test to assess the saccular and inferior vestibular nerve function
Ocular Vestibular Evoked Myogenic Potential Testing | baseline
  A vestibular function test to assess the utricular and superior vestibular nerve function
Ocular Motor Testing | baseline
  A vestibular function test to evaluate oculomotor function
Dix-Hallpike Test | baseline
  A diagnostic maneuver to identify benign paroxysmal positional vertigo
Roll Test | baseline
  A diagnostic maneuver to identify benign paroxysmal positional vertigo
Static visual acuity | baseline
  Static visual acuity measured using a Snellen chart (static logMAR)
Dynamic visual acuity | baseline
  Visual acuity during head movement measured using a Snellen chart relative to static visual acuity (static logMAR - dynamic logMAR)
Dizziness Handicap Inventory | baseline
  A 25-item self-assessment inventory to evaluate self-perceived handicapping effects of dizziness (0-100). Higher scores indicate a greater perceived handicap due to dizziness.

OTHER OUTCOMES:
Age | baseline
  Years since birth
Sex | baseline
  Male or female
Montreal Cognitive Assessment | baseline
  A screening test to assess global cognition (0-30). Higher scores indicate better performance.
Shortened Iconographical Falls Efficacy Scale | baseline
  A 10-item scale to assess fear of falling. Each item is scored on a 4-point scale (1 = not at all concerned to 4 = very concerned).
Fall history | baseline
  Number of falls in the past month
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part I | baseline
  A 13-item rating scale to assess non-motor experiences of daily living (0-52). Higher scores indicate a worse outcome.
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III | baseline
  An 18-item motor examination to assess motor symptoms (0-132). Higher scores indicate a worse outcome.
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part IV | baseline
  A 6-item rating scale to assess motor complications. Higher scores indicate a worse outcome.
Hoehn and Yahr scale | baseline
  A scale to assess disease severity/progression (0-5). Higher scores indicate more severe symptoms.
New Freezing of Gait Questionnaire | baseline
  A 9-item questionnaire to assess freezing of gait severity (0-28). Higher scores indicate more severe freezing of gait.
Time since diagnosis | baseline
  The number of days since the diagnosis of Parkinson's Disease
Blood pressure | baseline
  The ratio of systolic over diastolic blood pressure (mm Hg)
Medication | baseline
  Number, type and dose (mg) of medication

CONTACTS AND LOCATIONS:
Overall Officials: Katie Bouche, PhD, Principal Investigator — University Hospital, Ghent; Leen Maes, PhD, Principal Investigator — University Ghent; Anke Van Bladel, PhD, Principal Investigator — University Ghent; Nina Lefeber, PhD, Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - Ghent University Hospital, Ghent
  - Ghent University, Ghent